CLINICAL TRIAL: NCT01990729
Title: Efficacy and Safety of ARTRA (Glucosamine Plus Chondroitin Sulfate Combination) in Treatment of Non-specific Chronic Low Back Pain of Lumbosacral Localization in Ambulatory Care
Brief Title: Efficacy and Safety of ARTRA (Glucosamine Plus Chondroitin Sulfate Combination) in Treatment of Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Unipharm, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARTRA-PMS-LBP/2012
Record Dates: First submitted 2013-10-07; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — hydroquinone; Glucosamine; Chondroitin Sulfates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARTRA: Patients with low back pain treated with ARTRA.
  Interventions: Dietary Supplement: ARTRA

INTERVENTIONS:
Dietary Supplement: ARTRA — ARTRA (glucosamine and chondroitin sulfate)
  Other Names: Glucosamine; Chondroitin sulfate

SUMMARY:
To study the safety and efficacy of ARTRA (glucosamine chondroitin sulfate) in the treatment of non-specific low-back pain of lumbosacral localization in ambulatory care.

DETAILED DESCRIPTION:
We enrolled patients between 40 and 65 years of age who had low back pain for at least 12 weeks with a pain intensity >3 on a 0-10 point visual analogue scale (VAS). Major exclusion criteria were presence of fibromyalgia, degenerative spondylolisthesis, and alcohol and/or drug abuse. All patients were treated with ARTRA (combination of glucosamine hydrochloride 500 mg and chondroitin sulfate 500 mg in tab; Unipharm Inc.) at a dose of 1 tab bid for the first month and then 1 tab daily for the next two months. The primary endpoint was pain intensity (at rest and movement) as measured on a 0-10 point VAS. Secondary endpoints included Oswestry Disability Index, patient global assessment of efficacy (0-5 scale) and NSAID consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 40-65 years, inclusively.
2. Pain intensity according to Visual Analogue Scale (VAS) > 3 points.
3. Duration of back pain > 12 weeks.
4. Pain reinforcement during movement in lumbar spine.
5. Osteoarthritis, spondylarthrosis, osteochondrosis.
6. Given written Informed consent form for participation in the study.
7. Treatment with ARTRA

Exclusion Criteria:

1. History of allergic reactions to chondroprotectors.
2. Participation in another clinical study within 30 days before screening or during this study.
3. Fibromyalgia.
4. Active neoplastic disease, history of neoplastic disease within 3 years before screening.
5. Paget's disease.
6. Degenerative spondylolisthesis.
7. Administration of anticonvulsant, antidepressant, barbiturate, anxiolytic, or muscle relaxant drugs for more than one week prior screening.
8. History of alcohol or drug abuse.
9. Frequent episodes of nausea, dyspepsia, pain in the epigastric region, diarrhea, face and extremities edema, dizziness and headache.
10. History of any disease that, in the opinion of the investigator, might confound the results of the study or poses an additional risk to the subject during participation in the study
11. Clinically significant renal disorders.

    -

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain in ambulatory care
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 3 months
  Pain intensity on Visual Analogue Scale

SECONDARY OUTCOMES:
Oswestry Disability Index | 3 months
Patient global assessment of efficacy | 3 months
NSAID consumption | 3 months
  Number of patients taking NSAIDs

CONTACTS AND LOCATIONS:
Overall Officials: Gurkirpal Singh, MD, Study Chair — Irish Clinical Outcomes in Research and Education
Locations (1):
- FGBU "State NII of Rheumatology" of RAMS, Moscow, Russia